CLINICAL TRIAL: NCT07381725
Title: A Comparative Analysis of Single Lateral Plate Versus Double Plating for the Fixation of Distal Femoral Fractures: A Randomized Clinical Trial
Brief Title: Single Lateral Plate Versus Double Plating for the Fixation of Distal Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelkader, Lecturer of Orthopedic Surgery, Faculty of Medicine, Beni-Suef University, Egypt., Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/02102022/Ali
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Single Lateral Plate; Double Plating; Fixation; Distal Femoral Fractures
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Single Plate): (Experimental): Patients underwent open Reduction and Internal Fixation (ORIF) using a single pre-contoured lateral distal femoral locking compression plate via a standard lateral approach.
  Interventions: Procedure: Single lateral distal femoral locking compression plate
- Group II (Double Plate) (Experimental): Patients underwent open Reduction and Internal Fixation (ORIF) using a lateral distal femoral locking plate combined with a medial buttress plate (3.5mm reconstruction plate) via an anterolateral approach with subvastus medial dissection.
  Interventions: Procedure: Double Plating

INTERVENTIONS:
Procedure: Single lateral distal femoral locking compression plate — Patients underwent open Reduction and Internal Fixation (ORIF) using a single pre-contoured lateral distal femoral locking compression plate via a standard lateral approach.
  Arms: Group I (Single Plate):
Procedure: Double Plating — Patients underwent open Reduction and Internal Fixation (ORIF) using a lateral distal femoral locking plate combined with a medial buttress plate (3.5mm reconstruction plate) via an anterolateral approach with subvastus medial dissection.
  Arms: Group II (Double Plate)

SUMMARY:
This trial aimed to provide Level I evidence on the comparative effectiveness, safety, and functional outcomes of single versus double plating for distal femoral fractures.

DETAILED DESCRIPTION:
Distal femoral fractures, particularly those with metaphyseal comminution, present a significant surgical challenge with high risks of nonunion, malalignment, and functional impairment.

The single lateral locking plate (SLP) is a common fixation method but may lack sufficient stability in complex fractures, leading to varus collapse.

Dual plating (lateral and medial plates) offers enhanced biomechanical stability but involves greater surgical invasiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Acute, displaced, closed or Gustilo-Anderson Type I open distal femoral fracture (AO/OTA types 33-A1, A2, A3, C1, C2, C3).
* Presentation within 7 days of injury.
* Provision of written informed consent.

Exclusion Criteria:

* Pathological fractures.
* Associated ipsilateral lower extremity trauma (floating knee).
* Associated neurovascular injury requiring repair.
* Pre-existing symptomatic knee arthritis or prior major knee surgery.
* Active local or systemic infection.
* Medical comorbidities precluding surgery or anesthesia [American Society of Anesthesiologists (ASA) class IV/V].
* Cognitive impairment or inability to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | 6 months post-surgery
  The Knee Society Score (KSS) contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.

SECONDARY OUTCOMES:
Radiological Union | 52 weeks post-surgery
  Radiological Union (defined as bridging callus in 3/4 cortices) was recorded. It was assessed at 2, 6, 12, 24, and 52 weeks post-surgery.
Active Range of Motion | 52 weeks post-surgery
  Active Range of Motion was measured with a goniometer assesses the joint angle achieved through a patient's voluntary muscle contraction, without external assistance. It was assessed at 2, 6, 12, 24, and 52 weeks post-surgery.
Degree of pain | 52 weeks post-surgery
  Degree of pain was assessed using Visual Analogue Scale (VAS). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). It was assessed at 2, 6, 12, 24, and 52 weeks post-surgery.
Fracture Alignment | 52 weeks post-surgery
  Fracture Alignment on Anterior Posterior (AP)/Lateral radiographs was recorded. It was assessed at 2, 6, 12, 24, and 52 weeks post-surgery.
Assessment of quality of Life | 12 months post-surgery
  Quality of Life was assessed using EQ-5D-5L questionnaire across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It was assessed at 6 and 12 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.